CLINICAL TRIAL: NCT05884866
Title: Natriuretic-ureothelic Adaptation of Body Fluid Homeostasis During SGLT-2 Inhibition and/or Mineralocorticoid Receptor Modulation in Patients With Chronic Kidney Disease. A 4-arm, Double-blind, Double-dummy, Parallel-group, Phase 2 Study to Investigate the Mechanistic Effects of Dapagliflozin, Dapagliflozin + Balcinrenone, Balcinrenone and Placebo on Body Solute and Water Homeostasis and Energy Metabolism in Male and Female Participants Over 50 Years of Age With Chronic Kidney Disease.
Brief Title: A Study to Investigate the Mechanistic Effects of Dapagliflozin Alone or in Combination With Balcinrenone, Compared to Balcinrenone and Placebo on Body Fluid and Electrolyte Handling and Energy Metabolism in Participants Over 50 Years of Age With Chronic Kidney Disease.
Acronym: DapaBalci-Leap
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Adriana Marton, Principal Investigator, Klinikum Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT114-2022-01; 2022-002721-99 (EudraCT Number)
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Chronic Renal Failure; Mechanistic Effects of SGLT2 Inhibition and/ or MR Antagonism on Body Fluid and Electrolyte Homeostatis; Chronic Kidney Disease Stage 3; Electrolyte and Fluid Balance Conditions
Keywords: Chronic kidney disease; Water conservation; SGLT2 inhibitors, dapagliflozin; MR antagonists, balcinrenone; Amino acids; Energy metabolism
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: 4-arm, double-blind, double-dummy, parallel-group
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dapagliflozin (Active Comparator): 1 tablet Dapagliflozin 10 mg + 1 capsule Balcinrenone 50mg matching Placebo + 1 capsule Balcinrenone 100 mg matching Placebo
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Balcinrenone 50mg matching Placebo; Drug: Balcinrenone 100mg matching Placebo
- Balcinrenone (Experimental): 1 capsule Balcinrenone 50mg + 1 capsule Balcinrenone 100 mg + 1 tablet Dapagliflozin matching Placebo
  Interventions: Drug: Balcinrenone 50mg Capsule; Drug: Balcinrenone 100mg Capsule; Drug: Dapagliflozin matching Placebo
- Dapagliflozin + Balcinrenone (Experimental): 1 tablet Dapagliflozin 10mg + 1 capsule Balcinrenone 50mg + 1 capsule Balcinrenone 100 mg
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Balcinrenone 50mg Capsule; Drug: Balcinrenone 100mg Capsule
- Placebo (Placebo Comparator): 1 tablet Dapagliflozin matching Placebo + 1 capsule Balcinrenone 50mg matching Placebo + 1 capsule Balcinrenone 100 mg matching Placebo
  Interventions: Drug: Dapagliflozin matching Placebo; Drug: Balcinrenone 50mg matching Placebo; Drug: Balcinrenone 100mg matching Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — see arms
  Other Names: Forxiga
  Arms: Dapagliflozin; Dapagliflozin + Balcinrenone
Drug: Balcinrenone 50mg Capsule — see arms
  Arms: Balcinrenone; Dapagliflozin + Balcinrenone
Drug: Balcinrenone 100mg Capsule — see arms
  Arms: Balcinrenone; Dapagliflozin + Balcinrenone
Drug: Dapagliflozin matching Placebo — see arms
  Arms: Balcinrenone; Placebo
Drug: Balcinrenone 50mg matching Placebo — see arms
  Arms: Dapagliflozin; Placebo
Drug: Balcinrenone 100mg matching Placebo — see arms
  Arms: Dapagliflozin; Placebo

SUMMARY:
The purpose of this study is to investigate the mechanistic effects of dapagliflozin 10 mg, alone or in combination with balcinrenone 150 mg, with balcinrenone 150 mg and placebo, on the way the body handles electrolytes and water content, as well as the effects these interventions may have on energy metabolism in participants with stage 3 chronic kidney disease.

The study interventions will be administered orally, daily, in addition to current therapy, for a duration of 28 days. This will allow us to maximize our ability to detect a drug effect while minimizing the drop-out rate that accompanies longer studies.

In order to understand the different mechanistic effects of these interventions on energy metabolism, the study will be conducted at two study sites. The study design and treatment allocation, treatment duration as well as sample analysis for evaluation of the primary endpoint will be identical for all participants, at both sites. Therefore, urine and plasma samples for analysis of water and electrolyte handling will be collected from all study participants at both sites.

In addition to the primary endpoint, the main study site (Nuremberg) will conduct a metabolic study to investigate the early- and late-effects of the interventions, while the second site, Marseille, will conduct an imaging sub-study to assess changes at the tissue level before and after treatment.

DETAILED DESCRIPTION:
The Nuremberg site will perform metabolomics analyses and evaluation of metabolic longevity switches in erythrocytes; participants will be randomly allocated to 1 of the 4 treatment arms, with n=25 participants per arm.

All participants in Nuremberg will undergo 3 study visits: at baseline, day 3 (to study the early effect of the intervention) and at day 28 (for the late metabolic effects). An additional safety study visit will take place at day 7+/-1. A follow-up visit will take place at day 28 +/- 7 after the last dose.

Study procedures: medical examination, height, weight, blood pressure (BP), heart rate (HR), 24h urine collection and analysis, venous blood sampling.

This site will prepare venous blood samples for metabolomic analysis and will perform the erythrocyte isolation protocol for the assessment of erythrocyte metabolism.

The Marseille site will conduct an imaging sub-study to evaluate tissue sodium and water content, and muscle energy metabolism before and after the study intervention; participants will be randomly allocated to 1 of the 4 treatment arms, with n=10 participants per arm.

All participants in Marseille will undergo 2 study visits: at baseline (before starting the intervention) and after 28 days of treatment. An additional safety study visit will take place at day 7+/-1. A follow-up visit will take place at day 28 +/- 7 after the last dose.

Study procedures: medical examination, height, weight, blood pressure, heart rate, 24h urine collection and analysis, venous blood sampling, MRI scans.

During each of the study visits at baseline and day 28 the participants will undergo 2 MRI scans: a 23Na MRI scan for the assessment of tissue sodium storage and water content at ultra-high field (7T MRI) and a spectroscopy scan for the assessment of muscle energy metabolism (phosphorus spectroscopy at 3T). The total duration of the scans at each study visit will be approximately 2h.

The Marseille recruitment site has been closed in October 2024 because of low recruitment rate. The recruitment will be completed in Nuremberg, and the number of patients has been increased to 25 patients per arm. Considering the very low drop-out rate in Nuremberg (2%) a total of 100 participants (25 per arm) will be randomized into the study. This number will suffice to achieve the necessary sample size of 23 patients for arm, and meet the necessary sample size for the primary endpoint according to the initial statistical power calculation : 23 per arm, accounting for a drop-out rate of 8%.

Enrolled means participants' or their legally acceptable representatives' agreement to participate in a clinical study following completion of the informed consent process. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening.

Participants in this study will be randomized into one of the 4 treatment arms:

1. Balcinrenone 150 mg (n=30)
2. Balcinrenone 150 mg + Dapagliflozin 10 mg (n=30)
3. Dapagliflozin 10 mg (n=30)
4. Placebo (n=30) For each group, 25 participants per group will complete the study (total n=100).

No dose modification, neither for dapagliflozin nor for balcinrenone, is planned during this study. To ensure a dose interval of about 24 hours, the medication should be taken every day in the morning. If a dose is missed by more than 12 hours, that dose should be skipped and the next dose should be taken as scheduled. No double doses should be taken.

Because of the short treatment duration in this study (28 days) no temporary discontinuation can take place, as this can affect the metabolic phenotype at day 3 and day 28. Therefore, if a participant needs to discontinue the study intervention, this participant will be withdrawn from the study and replaced.

Treatment duration will be 28 days, up to a maximum of 32 days to allow for scheduling flexibility. A follow-up visit will take place approximately one month (28 days +/-7 days) after the end of the intervention period. The screening visit may take place anytime within 4 weeks prior to Baseline visit. Therefore, the estimated total study duration for each participant, including screening and follow-up is 2 to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic kidney disease, with eGFR ≥30 and ≤60 mL/min/1.73m2
* Serum/ plasma K+ levels ≥ 3.5 and < 5.0 mmol/L OR within normal laboratory ranges when these are provided, within 2 weeks prior to randomization
* Serum/plasma Na+ levels within normal reference values within 2 weeks prior to randomization
* If participants have type 2 diabetes mellitus, treatment with metformin, sulphonylureas, DPP4 inhibitors or any combinations of these agents with or without insulin would be accepted but is not mandatory. If used, stable dose of metformin, sulphonylureas, or DPP4 inhibitors or their combination as anti-diabetic therapy for the 12 weeks prior to randomization is required
* No changes in background treatment for at least 3 weeks prior to randomization
* Body mass index less than 40 kg/m2
* Negative pregnancy test (urine or serum) for female subjects of childbearing potential and willingness to use a highly effective birth control (see Appendix 4) if of childbearing potential.
* Willingness to participate and ability to provide signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Uncontrolled type 2 diabetes mellitus with HbA1C > 10.5% in the most recent medical records
* Participants with type 2 diabetes mellitus treated with insulin if insulin dosing (intermediate, long-acting, premixed insulin, basal bolus insulin) was not stable in the 12 weeks prior to randomization as judged by the Investigator
* Patients with systolic blood pressure levels <100 mmHg at the time of enrolment
* Patients with congestive heart failure NYHA stage IV or hospitalized for decompensation of heart failure in the 3 months prior to screening
* History of any life-threatening cardiac arrhythmias, or uncontrolled ventricular rate in participants with atrial fibrillation or atrial flutter
* Acute coronary syndrome and/or percutaneous cardiac interventions within 3 months prior to screening
* Unstable or rapidly progressing renal disease
* Chronic cystitis and recurrent genital or urinary tract infections
* Significant hepatic disease, including hepatitis and/or liver cirrhosis (Child-Pugh class A-C), or AST or ALT > 2 × ULN (upper limit of normal); or total bilirubin levels (TBL) > 2 × ULN; or serum albumin levels < 3.5 g/dL
* Medical conditions associated with development of hyperkalemia (Addison's disease)
* Stroke, transient ischemic attack, carotid surgery, or carotid angioplasty within 3 months prior to screening
* Hemoglobin levels below 8.5 g/dL or over 15 g/dL OR over the normal laboratory ranges, when these are provided
* Patients who have received an organ transplant at any time or bone marrow transplant in the previous 10 years
* HIV infection
* Active cancer, history of bladder cancer
* Patients who have had major surgery in the 3 months prior to screening
* Patients with muscular dystrophies
* Patients who have severe comorbid conditions likely to compromise survival or study participation
* Pregnant and breast-feeding women
* Medical treatment with either a mineralocorticoid receptor antagonist (MRA) or a sodium-glucose co-transporter-2 inhibitor (SGLT2i) within 3 months prior to screening
* Medical treatment with potassium binders
* Medical treatment with strong or moderate CYP3A4 inducers or inhibitors
* Prior serious hypersensitivity reaction to dapagliflozin (Forxiga®), balcinrenone or to any of their excipients
* Treatment with cytotoxic therapy, immunosuppressive therapy or other immunotherapy within 6 months prior to screening
* Unwillingness or other inability to cooperate
* For patients undergoing MRI scans, presence of implanted devices (surgical clips, heart pacemakers or defibrillators, cochlear implants), iron-based tattoos, any other pieces of metal or devices that are not MR-safe anywhere in the body

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To show that treatment with balcinrenone preserves the beneficial dapagliflozin-driven increase in 24h renal glucose excretion | 28 days
  Change from baseline in 24h urine glucose excretion at day 28

SECONDARY OUTCOMES:
To demonstrate that the dapagliflozin induced increase in urine solute concentration is not altered by balcinrenone | 28 days
  Change from baseline in urine osmolality at day 3 and day 28
To demonstrate that treatment with dapagliflozin, with or without balcinrenone reduces free-water clearance within 48h, and further urine concentration is observed after 4 weeks | 28 days
  Change from baseline in free water clearance at day 3 and day 28
To demonstrate that treatment with dapagliflozin, with or without balcinrenone, increases the contribution of glucose to osmoticdiuretic volume formation within 48h, and that this effect persists after 4 weeks | 28 days
  Change from baseline in urine glucose fraction at day 3 and day 28
To demonstrate that treatment with dapagliflozin, with or without balcinrenone, decreases the contribution of sodium and urea to osmotic-diuretic volume formation within 48h, and that this effect persists after 4 weeks | 28 days
  Change from baseline in urine sodium fraction at day 3 and day 28; Change from baseline in urine urea fraction at day 3 and day 28
To demonstrate that treatment with dapagliflozin, with or without balcinrenone, does not change the contribution of potassium to osmotic-diuretic volume formation within 48h, and that this effect persists after 4 weeks | 28 days
  Change from baseline in urine potassium fraction at day 3 and day 28
To demonstrate that treatment with dapagliflozin with or without balcinrenone does not change body water content after 4 weeks | 28 days
  Change from baseline in muscle water content as measured at 7T MRI at day 28
To demonstrate that patients treated with dapagliflozin alone or in combination with balcinrenone show increased plasma copeptin levels within 48h and/or after 4 weeks | 28 days
  Change from baseline in copeptin levels at day 3 and day 28
To demonstrate that patients treated with dapagliflozin alone or in combination balcinrenone show increased plasma glucagon and reduced plasma insulin levels within 48h and/or after 4 weeks | 28 days
  Change from baseline in plasma insulin/glucagon ratio at day 3 and day 28

OTHER OUTCOMES:
To demonstrate that treatment with dapagliflozin and/or balcinrenone for 4 weeks does not change tissue Na+ content as measured with MRI at 7T | 28 days
  Change from baseline in tissue Na+ content at day 28
To demonstrate that treatment with dapagliflozin with or without balcinrenone will increase muscle nitrogen transfer and induce pH changes during the rest-exercise-recovery period | 28 days
  Change from baseline in pH levels levels at day 28 as quantified with 31P spectroscopy at 3T MRI
To test the hypothesis that parallel to RAAS activation, patients treated with dapagliflozin show increased 24h urine cortisol excretion independent of parallel balcinrenone treatment | 28 days
  Change from baseline in 24h urine cortisol levels at day 3 and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Marton, MD, Principal Investigator — Klinikum Nuernberg
Locations (2):
- Assistance Publique-Hopitaux de Marseille (AP-HM), Marseille, France
- Klinikum Nuernberg, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data (IPD) collected during study visits will be shared, and only for participants who have provided informed consent for data sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2 years after article publication with no end date
Access Criteria: Access will be granted upon reasonable request, provided that interested researchers have a scientific hypothesis for which they submit a methodologically sound proposal, including clearly defined research hypothesis and a statistical analysis plan. To gain access, data requesters must comply with applicable ethical and data protection regulations. Proposals should be directed to the Principal Investigator (Adriana Marton) and/or Data Manager (Jens Titze) via email.

REFERENCES:
- [Background] Marton A, Kaneko T, Kovalik JP, Yasui A, Nishiyama A, Kitada K, Titze J. Organ protection by SGLT2 inhibitors: role of metabolic energy and water conservation. Nat Rev Nephrol. 2021 Jan;17(1):65-77. doi: 10.1038/s41581-020-00350-x. Epub 2020 Oct 1. PMID 33005037
- [Background] Kovarik JJ, Morisawa N, Wild J, Marton A, Takase-Minegishi K, Minegishi S, Daub S, Sands JM, Klein JD, Bailey JL, Kovalik JP, Rauh M, Karbach S, Hilgers KF, Luft F, Nishiyama A, Nakano D, Kitada K, Titze J. Adaptive physiological water conservation explains hypertension and muscle catabolism in experimental chronic renal failure. Acta Physiol (Oxf). 2021 May;232(1):e13629. doi: 10.1111/apha.13629. Epub 2021 Mar 7. PMID 33590667
- [Background] Wild J, Jung R, Knopp T, Efentakis P, Benaki D, Grill A, Wegner J, Molitor M, Garlapati V, Rakova N, Marko L, Marton A, Mikros E, Munzel T, Kossmann S, Rauh M, Nakano D, Kitada K, Luft F, Waisman A, Wenzel P, Titze J, Karbach S. Aestivation motifs explain hypertension and muscle mass loss in mice with psoriatic skin barrier defect. Acta Physiol (Oxf). 2021 May;232(1):e13628. doi: 10.1111/apha.13628. Epub 2021 Feb 23. PMID 33590724
- [Background] Kitada K, Daub S, Zhang Y, Klein JD, Nakano D, Pedchenko T, Lantier L, LaRocque LM, Marton A, Neubert P, Schroder A, Rakova N, Jantsch J, Dikalova AE, Dikalov SI, Harrison DG, Muller DN, Nishiyama A, Rauh M, Harris RC, Luft FC, Wassermann DH, Sands JM, Titze J. High salt intake reprioritizes osmolyte and energy metabolism for body fluid conservation. J Clin Invest. 2017 May 1;127(5):1944-1959. doi: 10.1172/JCI88532. Epub 2017 Apr 17. PMID 28414295